CLINICAL TRIAL: NCT06047054
Title: Incidence Rate and Risk Factors of Malnutrition in Patients Admitted to Surgical Intensive Care Unit
Brief Title: Incidence Rate and Risk Factors of Malnutrition in ICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Naglaa Fathy Abdelhaleem Abdelhaleem, lecturer of anesthesia and ICU, Zagazig University
Other Study IDs: IRB #7074
Record Dates: First submitted 2023-08-30; First posted 2023-09-21 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2023-08

CONDITIONS: Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess the incidence of malnutrition in surgical Intensive Care Unit by NUTRIC score. To determine the different risk factors of malnutrition

DETAILED DESCRIPTION:
To assess the incidence of malnutrition in surgical Intensive Care Unit by NUTRIC score. To determine the different risk factors of malnutrition by assessment of the type of nutrition, caloric adequacy, and actual caloric intake, laboratory Investigations twice weekly

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who will be admitted to surgical ICU.
* Both sexes.

Exclusion Criteria:

* • Referral from another hospital or other ICU

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All cases who will admitted to the surgical intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Assess incidence rate of malnutrition in ICU | From the date of randomization until the date of ICU discharge or death, assessed up to 4 months
  Assessment of nutrition state by (NUTRIC) Score on admission and weekly until patient discharge or death

SECONDARY OUTCOMES:
Correlation of risk factors with malnutrition in ICU | From the date of randomization until the date of ICU discharge or death, assessed up to 4 months
  correlation of risk factors such as: age, comorbidities, and sepsis with malnutrition

CONTACTS AND LOCATIONS:
Overall Officials: Naglaa Abdelhaleem, MD, Principal Investigator — Faculty of medicine, Zagazig University Hospitals
Locations (1):
- Faculty of Medicine - Zagazig University, Zagazig, Egypt

REFERENCES:
- [Background] Lew CCH, Yandell R, Fraser RJL, Chua AP, Chong MFF, Miller M. Association Between Malnutrition and Clinical Outcomes in the Intensive Care Unit: A Systematic Review [Formula: see text]. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):744-758. doi: 10.1177/0148607115625638. Epub 2016 Feb 2. PMID 26838530